CLINICAL TRIAL: NCT02212210
Title: Maternal Epidural Steroids to Prevent Neonatal Exposure to Hyperthermia and Inflammation
Brief Title: Maternal Epidural Steroids and Hyperthemia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI permanently closed accrual for the study based on FDA warning issued in April 2014. Study is closed
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christopher G. Goodier, Instructor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Goodier_Epidural_Steroids
Record Dates: First submitted 2014-08-04; First posted 2014-08-08 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2014-08

CONDITIONS: Fever; Labor Pain; Complication of Anesthesia During Pregnancy, Unspecified
MeSH Terms: conditions — Fever; Labor Pain | interventions — Methylprednisolone; Methylprednisolone Acetate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): 1cc of 80mg methylprednisolone to be diluted with 1cc preservative free normal saline
  Interventions: Drug: Methylprednisolone
- Normal saline (Placebo Comparator): 2cc preservative free normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Methylprednisolone
  Other Names: DEPO-MEDROL
  Arms: Methylprednisolone
Drug: Normal saline
  Other Names: Saline placebo
  Arms: Normal saline

SUMMARY:
The purpose of this study is to look to see if adding steroids to an epidural reduces the chances of having a fever in labor, and protects the baby from exposure to inflammation.

DETAILED DESCRIPTION:
The association between epidural analgesia and increased maternal intrapartum temperature has been well documented in multiple randomized controlled trials. The exact mechanism for this elevation in temperature is unknown; however the most likely cause appears to be non-infectious inflammatory stimulation. Fetal exposure to maternal fever in utero has been linked with increased antibiotic treatment, increased neonatal sepsis evaluation, and longer length of stay for neonates. In addition there is evidence to suggest intrapartum fevers may lower the threshold for fetal hypoxic brain injury and increase the risk of cerebral palsy. The risk of neonatal encephalopathy in infants born to febrile mothers is 1% compared to 0.1% to afebrile mothers. Safe interventions are needed to prevent adverse fetal outcomes.

ELIGIBILITY:
Inclusion criteria:

* Nulliparity
* Age>=18
* Patient requests epidural analgesia
* GA >= 37 weeks

Exclusion criteria:

* No prenatal care
* Temperature >99.4 at decision for epidural placement
* Cervical dilation >4cm
* Diabetes (pre-gestational or gestational)
* Autoimmune condition
* Pre-eclampsia
* Maternal heart disease
* Current steroid use
* Active infection (bacterial or viral)
* Wet Tap (CSF on placement of epidural)
* Pre-gestational diabetes
* Known systemic infection (bacterial, viral, fungal or tubercular)
* Known allergy to steroids
* Heart failure
* Hypertensive crisis
* History of active epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of maternal fever | delivery
  Oral maternal temperature will be collected hourly starting at epidural placement. Temperature will be recorded until delivery.

SECONDARY OUTCOMES:
Rate of funisitis | delivery
  Cord segment will be collected at time of delivery and fetal end identified and sent to pathologist for evidence of funisitis, grade and stage.

OTHER OUTCOMES:
IL-6 level | delivery
  Cord blood will be obtained at delivery and plasma will be assessed for IL-^ levels by standard ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Goodier, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States